CLINICAL TRIAL: NCT05633355
Title: A Phase 3, Open-label, 52-week Study to Assess the Safety, Tolerability, and Efficacy of Rocatinlimab (AMG 451) in Adolescent Subjects Aged ≥ 12 to < 18 Years With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-Orbit)
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of Rocatinlimab in Adolescent Participants With Moderate-to-severe Atopic Dermatitis (AD)
Acronym: ROCKET-Orbit
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210263; 2022-001548-99 (EudraCT Number)
Record Dates: First submitted 2022-11-22; First posted 2022-12-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Rocatinlimab; AMG 451; KHK4083
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rocatinlimab (Experimental): Rocatinlimab will be administered subcutaneously every 4 weeks (Q4W) for 52 weeks with one additional dose at Week 2.
  Interventions: Drug: Rocatinlimab

INTERVENTIONS:
Drug: Rocatinlimab — Subcutaneous (SC) injection
  Other Names: AMG 451

SUMMARY:
The primary objective of this study is to describe the safety and tolerability of rocatinlimab in adolescents with moderate-to-severe AD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 to < 18 years at day 1.
* Participant has a diagnosis of AD (according to American Academy of Dermatology Consensus Criteria [Eichenfield, 2014]) that has been present for at least 12 months before signing of informed consent
* Prior to informed consent, history of inadequate response to topical corticosteroids (TCS) of medium to higher potency (with or without topical calcineurin inhibitors [TCI] as appropriate) or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks)
* Eczema Area and Severity Index (EASI) score ≥ 12
* vIGA-AD score ≥ 3
* ≥ 10% BSA of AD involvement at day 1 pre-enrollment

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  * Systemic corticosteroids
  * Systemic immunosuppressants
  * Phototherapy
  * Oral or topical janus kinase inhibitors
* Treatment with any of the following agents within 1 week before day 1 pre-enrollment:

  * Topical PDE4 inhibitors
  * Other topical immunosuppressive agents (not including TCS/TCI)
  * Combination topical agents containing a high- or super-high potency corticosteroid

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Serious Adverse Events | Up to 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (77):
- United States (22):
  - Phoenix Childrens Hosptial, Phoenix, Arizona
  - Medical Advancement Centers of Arizona, Tempe, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Little Rock Allergy and Asthma Clinical Research Center, Little Rock, Arkansas
  - University of California Irvine, Irvine, California
  - University of California Los Angeles, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Manlio Dermatology, Kissimmee, Florida
  - Palm Springs Community Health Center, Miami, Florida
  - ARA Professionals Limited Liability Corporation, Miami, Florida
  - Deluxe Health Care LLC, Miami Lakes, Florida
  - Bluegrass Allergy Care, Lexington, Kentucky
  - Windsor Dermatology dba Eczema Treatment Center of New Jersey, East Windsor, New Jersey
  - Smart Medical Research Inc, Jackson Heights, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Auni Allergy, Findlay, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - DermDox Dermatology, LLC, Sugarloaf, Pennsylvania
  - Driscoll Childrens Hospital, Corpus Christi, Texas
  - Modern Research Associates, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - University of Utah MidValley Dermatology, Murray, Utah
- Argentina (6):
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Fundacion Cidea, Buenos Aires, Distrito Federal
  - Instituto de Neumonologia y Dermatologia, Buenos Aires, Distrito Federal
  - Centro de Investigaciones Clinicas Instituto Especialidades De La Salud De Rosario, Rosario, Santa Fe Province
  - Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Diagnostico ABC, Rosario, Santa Fe Province
- Australia (9):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - The Skin Hospital, Darlinghurst, New South Wales
  - Premier Specialists, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Monash Childrens Hospital, Clayton, Victoria
  - Institute for Skin Health and Immunity, Mitcham, Victoria
- Brazil (6):
  - Universidade Federal do Parana, Curitiba, Paraná
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Fundacao Abc - Centro Univ Fmabc, Santo André, São Paulo
  - Ispem-Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo, São Paulo
  - Alergoalfa Nucleo Diagnostico Tratamento e Pesquisa Clinica em Alergia, São Paulo
- Canada (13):
  - Dermatology Research Institute Incorporated, Calgary, Alberta
  - Stratica Dermatology, Edmonton, Alberta
  - Vida Clinical Research, Edmonton, Alberta
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - Skincare Studio, St. John's, Newfoundland and Labrador
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Halton Pediatric Allergy, Burlington, Ontario
  - LEADER Research, Hamilton, Ontario
  - Triple A Lab, Hamilton, Ontario
  - JRB Research Incorporated, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Toronto Research Centre Inc, Toronto, Ontario
  - FACET Dermatology, Toronto, Ontario
- University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (9):
  - Korea University Ansan Hospital, Ansansi, Gyeonggido
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - National Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
- Turkey (Türkiye) (5):
  - Bezmialem Vakif Universitesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bakircay Universitesi Cigli Egitim ve Arastirma Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (6):
  - Bristol Royal Hospital for Children, Bristol
  - Velocity Clinical Research, High Wycombe, High Wycombe
  - Alder Hey Childrens Hospital, Liverpool
  - Whipps Cross University Hospital, London
  - St Thomas Hospital, London
  - Carn to Coast Health Centres, Redruth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com